CLINICAL TRIAL: NCT03037125
Title: The Evaluation Of Bone Width Gain Following Split Crest Technique With Or Without PRF In Conjunction With Simultaneous Implant Placement In Narrow Alveolar Ridges: A Randomized Controlled Clinical Trial
Brief Title: The Evaluation Of Bone Width Gain Following Split Crest Technique With Or Without Platelet Rich Fibrin( PRF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Youssef Emad Zaghloul Meshreky, Bachelor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PERIO 3:7:3
Record Dates: First submitted 2017-01-19; First posted 2017-01-31 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Ridge Deficiency
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Split crest without PRF
  Interventions: Procedure: Split Crest without PRF
- Intervention Arm (Experimental): Split crest with PRF
  Interventions: Procedure: Split Crest with PRF

INTERVENTIONS:
Procedure: Split Crest with PRF — Narrow ridges are split to increase the ridge width and immediate implants are placed with PRF closing the gap
  Arms: Intervention Arm
Procedure: Split Crest without PRF — Narrow ridges are split to increase the ridge width and immediate implants are placed without grafting
  Arms: Control Arm

SUMMARY:
Split crest technique is a technique for horizontal bone augmentation used in case of narrow alveolar ridges as an alternative to the more aggressive techniques such as onlay bone grafting, guided bone regeneration (GBR) and distraction osteogenesis

The study goal is to evaluate whether if there will be any benefit of using platelet rich fibrin (PRF) with the split crest technique regarding bone width gain and healing response in comparison with split crest technique alone, where PRF is considered an autologous, growth factor containing material which is easy to collect and is of low cost.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with at least one missing tooth in the maxillary region
2. All the selected patients have a bucco-palatal width of the edentulous alveolar ridge from 3.5-5.5mm.
3. All the selected patients have at least 12 mm residual bone height at the edentulous area
4. The recipient site of the implant should be free from any pathological conditions.
5. No diagnosed bone disease or medication known to affect bone metabolism.
6. Patients who are cooperative, motivated, and hygiene conscious.

Exclusion Criteria:

1. Patients unable to undergo minor oral surgical procedures.
2. Patients with a history of drug abuse or catabolic drugs.
3. Patients with a history of psychiatric disorder.
4. Patients with unrealistic expectations about the esthetic outcome of implant therapy.
5. Patients with insufficient vertical inter-arch space, upon centric occlusion, to accommodate the available restorative components.
6. Patients in the growth stage with partially erupted teeth.
7. Patients who have any systemic condition that may contraindicate implant therapy.
8. Patients who have any habits that might jeopardize the osseointegration process, such as smoking and alcoholism.
9. Patients with parafunctional habits that produce overload on the implant, such as bruxism and clenching.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Bone width gain | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral and dental medicine, Cairo university, Cairo, Egypt